CLINICAL TRIAL: NCT04366869
Title: Which is More Effective in Management of Bruxism for Implant Overdenture Patients: Botox or Occlusal Splints - A One Year Clinical Study
Brief Title: Which is More Effective in Management of Bruxism: Botox or Occlusal Splints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Dina ElAwady, lecturer, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OctoberUMSA
Record Dates: First submitted 2020-04-21; First posted 2020-04-29 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Bruxism
MeSH Terms: conditions — Bruxism | interventions — Denture, Overlay; Occlusal Splints; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Active Comparator): traditional approach of removing denture at night
  Interventions: Device: overdenture
- intervention 1 (Experimental): occlusal splint
  Interventions: Device: occlusal splint
- intervention 2 (Experimental): Botox
  Interventions: Drug: Botox

INTERVENTIONS:
Device: overdenture — removal of overdenture at night
  Arms: control
Device: occlusal splint — occlusal splint on overdenture
  Arms: intervention 1
Drug: Botox — Botox injection i masseter in temporalis
  Other Names: Bolitinum Toxins
  Arms: intervention 2

SUMMARY:
The aim of this study is to compare the efficacy of Botulinum toxin (Botox) and traditional occlusal splints for the management of bruxism in edentulous patients rehabilitated with MIOD

DETAILED DESCRIPTION:
42 edentulous patients having implant retained mandibular overdenture suffering from bruxism with clinical manifestation, will be randomly divided into three groups, group 1 control group (traditional approach of removing denture at night) ,group 2 will be managed by occlusal splints whereas group 3 will be managed with botulinum toxin injection (Botox). New maxillary dentures and mandibular over dentures will be constructed for both groups. Muscle activity will be measured at time of denture insertion (T0), 3(T3) 6(T6), 9(T9) and 12(T12) month of treatment. Patients satisfaction will be evaluated at the time of denture insertion (T0), 6(T6), and 12(T12) month of treatment using TMD/ NS numeric scales 10 cm questionnaire which include: headache, face pain, face tension, limitation of mouth opening and complaints during mastication.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with bruxism
* patients had mandibular implant retained overdentures within the previous 3 years
* cooperative patients
* physically and psychologically able patients to tolerate the procedure

Exclusion Criteria:

* patients taking muscle relaxants
* patients without neuromuscular control
* poor oral hygiene

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction: questionnaire | 12months
  Patients satisfaction was evaluated using TMD/ NS numeric scales 10 cm questionnaire which included: headache, face pain, face tension, limitation of mouth opening and complaints during mastication with scores from 1 to 10 whereas 1 means least pain and 10 means highest pain.it was assessed at baseline (T0), then after 3months(T3) then after 6months from baseline(T6), then after 9months from baseline(T9) and finally after 12 months from baseline (T12). which means every 3 months.

SECONDARY OUTCOMES:
Electromyography | 12 months
  measuring muscle activity for massetter and temporalis muscle at baseline,3,6,9,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dina Elawady, PHD, Principal Investigator — Lecturer
Locations (1):
- MSA, Giza, Egypt